CLINICAL TRIAL: NCT02938468
Title: Efficacy and Safety of Dexamethasone in Management of Chronic Subdural Hematoma: A Single Center Randomized Control Trial
Brief Title: Mgt of Chronic Subdural Hematoma Using Dexamethasone
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB16-0219
Record Dates: First submitted 2016-09-21; First posted 2016-10-19 (Estimated); Last update posted 2020-07-01 (Actual); Status verified 2016-09

CONDITIONS: Chronic Subdural Hematoma
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery (Active Comparator): Patients in this arm will receive any form if surgical intervention (i.e. bedside burrhole craniostomy, 2 burrhole washout, craniotomy, endoscopy etc.) for treatment of their chronic subdural hematoma
  Interventions: Procedure: Any surgical intervention aim at treating chronic subdural hematoma
- Dexamethasone (Experimental): Patients in this arm will receive Dexamethasone over a 21day period for treatment of their chronic subdural hematoma
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone
  Other Names: Decadron
  Arms: Dexamethasone
Procedure: Any surgical intervention aim at treating chronic subdural hematoma
  Arms: Surgery

SUMMARY:
Chronic subdural hematoma (cSDH) is a collection of blood and its breakdown products in the subdural compartment. It is a condition frequently seen in any neurosurgical practice. cSDH is believed to arise from tearing of bridging veins as a result of trauma, which may be minor and unapparent to the patient. Management of cSDH is widely varied. A "wait-and-see" or "wait-and-rescan" approach may be acceptable in asymptomatic patients with a relatively small hematoma whilst cSDH with severe neurological deficits or decreased level of consciousness may require surgical decompression by burr-hole craniostomy, twist drill craniostomy or craniotomy. Surgery is associated with serious morbidity and mortality of up to 17% and recurrence rates of 4%-33% requiring further treatment in some instances.The safety and efficacy of different neurosurgical procedures have been evaluated but there is a paucity of well-designed randomized controlled trials in the literature. Consequently, there is no consensus on the best treatment with respect to surgical technique, pre-operative and post-operative management and nonsurgical alternatives including the use of Corticosteroids, Tranexamic acid, Osmotic diuretics, Atorvastatin or Angiotensin converting enzyme (ACE) inhibitors.

Corticosteroids may be a therapeutic option in the management of cSDH. There is very little data on the efficacy of corticosteroids in the treatment of cSDH and certainly no randomized trials. The purpose of the study is to prove dexamethasone can be just as efficacious as surgery in treating chronic subdural hematoma. The investigators also hope to show that those patients treated with dexamethasone suffer less complication compared to those who undergo surgery.

DETAILED DESCRIPTION:
Chronic subdural hematoma (cSDH) is a collection of blood and its breakdown products in the subdural compartment. It is a condition frequently seen in any neurosurgical practice. cSDH is believed to arise from tearing of bridging veins as a result of trauma, which may be minor and unapparent to the patient. The one-year incidence rate is 1 to 8.2 per 100 000 in those 65 years or older. Advanced age is one of several risk factors and the incidence is expected to increase due to improved life expectancy. Other risk factors include brain atrophy, chronic alcoholism, intracranial hypotension, male gender and coagulopathy (including antiplatelet and antithrombotic therapy).

Management of cSDH is widely varied. A "wait-and-see" or "wait-and-rescan" approach may be acceptable in asymptomatic patients with a relatively small hematoma whilst cSDH with severe neurological deficits or decreased level of consciousness may require surgical decompression by burr-hole craniostomy, twist drill craniostomy or craniotomy. Surgery is associated with serious morbidity and mortality of up to 17% and recurrence rates of 4%-33% requiring further treatment in some instances.The safety and efficacy of different neurosurgical procedures have been evaluated but there is a paucity of well-designed randomized controlled trials in the literature. Consequently, there is no consensus on the best treatment with respect to surgical technique, pre-operative and post-operative management and nonsurgical alternatives including the use of Corticosteroids, Tranexamic acid, Osmotic diuretics, Atorvastatin or Angiotensin converting enzyme (ACE) inhibitors.

Corticosteroids may be a therapeutic option in the management of cSDH. There is very little data on the efficacy of corticosteroids in the treatment of cSDH and certainly no randomized trials. The purpose of the study is to prove dexamethasone can be just as efficacious as surgery in treating chronic subdural hematoma. The investigators also hope to show that those patients treated with dexamethasone suffer less complication compared to those who undergo surgery.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 yrs
* subacute/chronic subdural hematoma on CT or MRI performed within 72 hours prior to recruitment
* patient must be symptomatic

Exclusion Criteria:

* Glasgow Coma Scale (GCS) ≤ 12
* patients needing craniotomy at the discretion of the on call neurosurgeon
* hemiparesis with less than antigravity (≤ 3/5 medical research council scale) strength in any testable myotomes

  °≥ 2 seizures at presentation or history of epilepsy
* subdural hematoma with an underlying lesion or condition such as tumor, arachnoid cyst, presence of a ventriculoperitoneal shunt or vascular malformation
* contraindication to dexamethasone including allergy or hypersensitivity to dexamethasone, immunocompromised/immunosuppressed patients, uncontrolled diabetes, untreated known peptic ulcer disease
* pregnant/breastfeeding mothers
* acute infection including latent/active tuberculosis (TB)
* history of psychosis
* anticoagulated for mechanical heart valve or arterial stent (i.e. coronary, carotid, or peripheral) placement
* small volume, non-operable subdural collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 326 (Estimated)
Dates: Start 2016-09-17 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Failure rates | 3 months
  Failure is defined as the requirement for surgical intervention in the dexamethasone group or re-operation in the surgical group.

SECONDARY OUTCOMES:
Recurrence rate | 3 months
  Recurrence is defined as symptomatic and radiologic re-accumulation of subdural hematoma on the ipsilateral side requiring a reoperation within 3months after treatment.
Modified Ranking Scale | 1, 3 and 6 months after treatment
  Functional outcome
Barthel index | 1, 3 and 6 months after treatment
  Functional outcome
Glasgow Outcome Scale | 1, 3 and 6 months after treatment
  Functional outcome
Glasgow Coma Scale | 1, 3 and 6 months after treatment
  Functional outcome
Markwalder score | 1, 3 and 6 months after treatment
  Functional outcome
Clinical improvement (Categorized as resolved, improved, unchanged or worse) | 1, 3 and 6 months after treatment
  Categorized as resolved, improved, unchanged or worse
Radiologic outcomes (Change in hematoma volume) | 1, 3 and 6 months after treatment
  Measured as change in hematoma volume
Quality of Life measured using the EQ-5D-5L | 1, 3 and 6 months after treatment
  Quality of life will be measured using the EuroQol health survey (EQ-5D-5L) questionnaire.
Mortality | 1, 3 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided